CLINICAL TRIAL: NCT05409261
Title: Phase II Trial Evaluating the Immunogenicity and Safety of Ad26.COV2.S Vaccine in Adult Participants in Mali
Brief Title: Evaluation of the Immunogenicity and Safety of Ad26.COV2.S's COVID-19 Vaccine
Acronym: CoviComMali
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: CEPI (Other); Innovative clinical research network in vaccinology (IREIVAC) (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); APHP (Other); Center for Vaccine Development - Mali (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ANRS0142S
Record Dates: First submitted 2022-04-01; First posted 2022-06-08 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; Vaccine Reaction; SARS CoV 2 Infection; Vaccine Adverse Reaction
Keywords: Ad26.COV2.S
MeSH Terms: conditions — COVID-19 | interventions — Ad26COVS1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ad26.COV2.S (Experimental): Single dose (0.5mL) of SARS-CoV-2 vaccine Ad26.COV2.S.
  Interventions: Biological: Ad26.COV2.S

INTERVENTIONS:
Biological: Ad26.COV2.S — Recombinant vaccine, contains Adenovirus type 26 encoding the SARS-CoV-2 spike glycoprotein
  Other Names: Janssen; Johnson&Johnson

SUMMARY:
Phase II, non-randomized, open-label, comparative, national, multicenter trial in Mali, aimed to assess the humoral vaccine immune response induced by Ad26.COV2.S vaccine in 200 adults one month after receiving the complete vaccination schedule of SARS-CoV-2 vaccine.

DETAILED DESCRIPTION:
The main objective of this phase II trial is to evaluate the humoral immune response induced by the Ad26.COV2.S vaccine in adults one month after complete vaccination regimen against SARS-CoV-2, compared younger (up to 45 years old) and elderly (55+ years old) populations.

200 participants will be included, 200 participants for each vacine. The age categories are 18 - 45 years, 55 - 64 years and 65+ years. The number of participants per age group will be distributed as follows 1:1:0,5. There will be no comparison between population on different vaccines.

Ad26.COV2 vaccine (200 participants) 18-45 years old, 80 participants 55-64 years old, 80 participants 65 years old or older, 40 participants

Participants in Ad26.COV2 arm receive intramuscularly as a single dose of 0.5mL.

Humoral vaccine immune responses, induced by Ad26.COV2.S vaccine, will be measured by ELISA at D0, M1, M2, M6, M12 and M24.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years old or 55 years and older
* Be eligible to receive one of the study vaccines as part of the trial
* Understand and agree to comply with study procedures (visits, telephone calls)
* Agree not to participate in any other vaccine study during the time of the study
* Give written informed consent prior to any examination performed as part of the trial

Exclusion Criteria:

* Positive SARS-CoV-2 antigenic test
* Positive SARS-CoV-2 polymerase chain reaction (PCR) results less than 48 hours old
* History of infection by SARS-CoV-2 confirmed by antigenic test or PCR within 3 months prior to inclusion
* Symptoms compatible with infection to SARS-CoV-2: sick or febrile participants (body temperature ≥ 38.0°C)
* Pregnant or breastfeeding woman
* Known chronic disease impacting the participant's immune response (uncured cancer, human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection)
* Anti-coagulant treatment
* Immunosuppressive treatment
* Contraindication to the proposed vaccine (according to RCP)
* Previously received at least one injection of a SARS-CoV-2 vaccine
* Patient having received immunoglobulin or another blood product within 3 months prior to inclusion
* A history of serious adverse vaccine reactions (anaphylaxis and associated symptoms such as rash, breathing difficulties, laryngeal edema, or a history of allergic reaction that may be exacerbated by a component of the SARS-CoV-2 vaccine)
* Any condition that, in the opinion of the investigator, may adversely affect the well-being of the participant and interfere with the purpose of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Anti-SARS-CoV-2 Spike immunoglobulin G (IgG) level | One month after complete vaccination schema
  Anti-SARS-CoV-2 Spike IgG level is measured using ELISA test

SECONDARY OUTCOMES:
Anti-SARS-CoV-2 Spike IgG level | At inclusion (Day 0) and then 1, 2, 6, 12, and 24 months after inclusion
  Anti-SARS-CoV-2 Spike IgG level is measured using ELISA test
Anti-SARS-CoV-2 immunoglobulin M (IgM) level | At inclusion (Day 0) and then 1, 2, 6, 12, and 24 months after inclusion
  Anti-SARS-CoV-2 IgM level is measured using ELISA test
Neutralizing antibody level for SARS-CoV-2 | Inclusion (Day 0) and then 1, 2, 6, 12, and 24 months after inclusion
  Neutralizing antibody levels specific for SARS-CoV-2 and its variants (conventional in vitro neutralization and pseudo-neutralization assays)
Fluorospot tests (type 1,2, and 17 helper T cell (TH1, TH2, TH17), Cytotoxicity) | Inclusion (Day 0) and then 2 and 6 months after inclusion
  Fluorospot tests (TH1, TH2, TH17, Cytotoxicity) Phenotyping of antigen-specific T cells by mass cytometry at Day 0 and Month 6 selected from the results of the Fluorospot test.
Mucosal SARS-CoV-2 specific antibody levels | Inclusion (Day 0) and then 1, 2, 6, 12, and 24 months after inclusion
  Mucosal SARS-CoV-2 specific antibody levels by measuring IgA, IgM and IgG in saliva using specific ELISAs
Determination of Epitope profile | Day 0 and Month 2
  Determination of epitope profile
B cell response to vaccine | Day 0, Month 2, Month 6
  Determination of repertoire of B cells (stereotype clonotype)
Measurement of ultrasensitive immunoglobulin A (IgA) and mucosal IgA and IgM functionality | Day 0 and then 1, 2, 6, 12, and 24 months after inclusion
  Measurement of ultrasensitive IgA in saliva by Photoring assay Measurement of mucosal IgA and IgM functionality by SARS-CoV-2 mucosal IgA- and IgM-specific antibody-dependent cell-mediated cytotoxicity (ADCC) test
Rate of adverse events | Between month 1 and month 24 after inclusion
  Rate of adverse events of any grade attributable to the vaccine or vaccination occurring between Month 1 and Month 24
SARS-CoV-2 infection | Date of inclusion until 24 months
  Occurrence of confirmed COVID-19 cases during participant follow-up

OTHER OUTCOMES:
Measurement of specific B memory cells and T cell response | B memory cells: Day 0 and then 2,6, and 12 months after inclusion., T cell : Inclusion (D0) and then at 12 months after inclusion
  Measurement of specific B memory cells (Elispot B) and T cell response (Cytof analysis)
Identification of predictive determinants of vaccine response | Day 0 until 24 months
  Identification of pre-existing immunity against other coronaviruses or respiratory pathogens, immunosenescence profile, transcriptomic, metabolomic and proteomic analysis, cytokine profile (IFNa), immune cell phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, Study Chair — Innovative clinical research network in vaccinology (I-REIVAC); Samba Sow, Principal Investigator — Center for Vaccine Development-Mali (CVD-Mali)
Locations (1):
- CVD-MALI, Bamako, Mali

IPD SHARING:
Plan to Share IPD: Yes